CLINICAL TRIAL: NCT05464056
Title: BUILT Family Lifestyle Program for Children with ADHD
Acronym: BUILT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: UIC Center for Health Equity Research (CHER) (Unknown); UIC Chicago Partnership for Health Promotion (CPHP) (Unknown); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Eduardo E. Bustamante, AssociateProfessor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0024
Record Dates: First submitted 2022-05-26; First posted 2022-07-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Lifestyle Intervention; Routines; Behavior change; Community-engaged research
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BUILT Study (Experimental): One group receives the intervention.
  Interventions: Behavioral: Be Unstoppable in Life Together (BUILT)

INTERVENTIONS:
Behavioral: Be Unstoppable in Life Together (BUILT) — Participants will complete weekly sleep, food, and exercise home challenges focused on creating sustainable healthy eating, sleep, and exercise routines. Parents will participate in weekly support calls by UIC and Chicago Park District staff to provide support and accountability. Children will have the opportunity to win small prizes based on completing weekly challenges. The intervention will be co-facilitated by UIC students and Chicago Park District staff and will largely take place on-line. For additional details visit: https://built.ahs.uic.edu.

SUMMARY:
The investigators have developed BUILT in hopes of empowering families to adopt and sustain healthy food, sleep, and exercise routines that optimize child focus, attention, and behavior. Over 6-weeks, the BUILT program will explore what science says about the effects of sleep, nutrition, and exercise on brain development and behavior; investigate the food, sleep, and exercise routines of the world's best athletes and intellectuals; and experiment with home routines to find those that best fits with participating families.

It is hypothesized that families participating in BUILT (N=150) will show significant improvements in child health behaviors (sleep, nutrition, physical activity, recreational screen time), child mental health (ADHD symptoms [primary outcome], child functional impairment), child physical literacy, and family dynamics (cohesion, structure, communication) from baseline to posttest.

DETAILED DESCRIPTION:
Families enrolled in Chicago Park District programs will be offered the opportunity to participate in the BUILT family lifestyle program. Using a single group design, measures will be taken within two weeks of program start and two weeks after completion. Additional feasibility measures will be taken during the program itself to inform refinements across iterations. The BUILT program will occur largely on-line and consist of weekly home challenges related to food, sleep, and exercise that add up to form a comprehensive home routine--the routine will optimize neurocognitive development and home structure. The program will be co-facilitated by UIC students and Chicago Park District staff. For more information visit the program website: https://built.ahs.uic.edu.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls ages 6 to 12 years old
* Parent orientation session summarizing activities
* Child free of conditions that preclude aerobic activity
* Child enrolled in Chicago Park District programming

Exclusion Criteria:

* Boys and girls < 6 years old or > 12 years old
* Parent does not participate in orientation session summarizing activities
* Child has conditions that preclude aerobic activity
* Child not enrolled in Chicago Park District programming

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 316 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Moderate-Vigorous Physical Activity at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Physical activity will be monitored for children at each time point with accelerometers worn at the wrist. Accelerometers provide a valid assessment of physical activity in free-living conditions. Data will be analyzed if ≥7 hours are available for ≥4 days. The outcome is minutes of moderate-vigorous physical activity per day and more minutes of moderate-vigorous physical activity are considered a better outcome.
Change from Baseline Sleep Quantity at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Sleep quantity will be monitored for children at each time point with accelerometers worn at the wrist. Accelerometers provide a valid assessment of sleep in free-living conditions. Sleep logs will differentiate sleep and wake times. More hours of sleep are considered a better outcome.
Change from Baseline Diet Quality at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Diet Quality will be assessed for each child at each time point using a Block Food Frequency Questionnaire (NutritionQuest). Higher scores on Diet Quality are considered a better outcome.
Change from Baseline Recreational Screen Time Quantity at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Recreational Screen time will be assessed by parent report of minutes of daily screen time on weekdays and weekends for school and non-school purposes, rounded to the nearest 15-minute increment. Fewer minutes of daily recreational screen time are considered a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Combined ADHD Symptoms at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Disruptive Behavior Disorder (DBD) Rating Scale lists the DSM-IV criteria for ADHD, ODD, and CD on a 4-point Likert scale from "not at all" to "very much." Each item is assigned a value (0 to 3) and these are summed to generate a continuous score on combined ADHD symptoms. Higher symptom scores are considered a worse outcome.
Change from Baseline Functional Impairment at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Impairment Rating Scale (IRS) assesses the severity of a child's impairment and need for treatment and services. Raters place an X on a line that signifies the child's placement on a continuum of impairment across seven domains. Under each domain rating is a section for the rater to describe his or her view of the child in a narrative. For scoring, the line is divided into seven equally spaced segments, and the segment where the X was placed constitutes the score between 0 (no problem/definitely does not need treatment or special services) and 6 (extreme problem/definitely needs treatment or special services). A 3 or above is scored as an impaired domain and these are summed as a continuous outcome. Higher numbers of domains endorsed as impaired are considered a worse outcome.
Change from Baseline Executive Function at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Behavioral Rating Inventory of Executive Function (BRIEF) assesses everyday manifestations of executive function. The tool consists of 86-items that use a scale from 0 "Never" to 2 "Often." The BRIEF generates a Global Executive Composite (GEC) score, which is standardized as a t-distribution where lower scores are considered a better outcome.
Change from Baseline Parental Stress at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Parental stress will be measured by the 10-item Perceived Stress Scale (PSS). Each item on the PSS uses a Likert scale ranging from 0 "Never" to 4 "Very Often." Higher scores on the PSS are considered a worse outcome.
Change from Baseline Home Structure at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Family Routines Inventory (FRI) is a 56-item questionnaire that divides routines into two pieces: the frequency of the routines and the importance of the routine. The frequency of the routine is recorded on a Likert scale from 0 "Almost Never" to 3 "Always Everyday." The importance of the routine is recorded on a Likert scale from 0 "Not at All Important" to 2 "Very Important." Overall higher frequency and importance scores are considered a better outcome.
Change from Baseline Family Cohesion at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Parenting and Family Adjustment Scale (PAFAS) is a brief measure of parental adjustment and parent-child relationship with good internal consistency and satisfactory construct and predictive validity. The PAFAS is a 30-item questionnaire that uses a 4-point scale from 0 (not at all) to 3 (very much). Subscales are summed into a family adjustment score where higher scores are considered a better outcome.
Change from Baseline Parent-Child Communication at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Parent-Child Communication will be measured with the Family Problem Solving Communication (FPSC) instrument, a 10-item measure of problem solving communication in families. A Likert scale is utilized for each statement and ranges from 0 "False" to 3 "True." A higher score on affirming communication and a lower score on incendiary communication are considered to be better outcomes.
Change from Baseline Physical Literacy at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Physical Literacy Assessment for Youth (PLAYfun) provides an assessment of key movement skills performed by children. The tool itself is made up of 18 tasks that cover the child's physical abilities. Each ability is graded on a four-point rubric with the following categories: Initial, Emerging, Competent and Proficient. Higher scores are considered to be a better outcome.
Change from Baseline Child Resilience at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  The Child and Youth Resilience Measure (CYRM-R) is a self-report measure of social-ecological resilience. This 17-item questionnaire uses a 5-point Likert scale that ranges from 0 "Not at All" to 4 "A Lot." Scores are summed and higher scores are considered a better outcome.
Change from Baseline Social Capital at Posttest | Baseline (within 2-weeks of intervention start date), Posttest (within 2-weeks of intervention end date)
  Social capital will be assessed by the 10-item Community Collective Efficacy (CCE) scale. The CCE uses a 5-point Likert scale ranging from 1 "Strongly Agree" to 5 "Strongly Disagree." Scores are summed and lower scores are considered a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo E Bustamante, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- Chicago Park District, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No